CLINICAL TRIAL: NCT03298165
Title: Diode Laser Cavity Disinfection (A Six Month Randomized Clinical Trial).
Brief Title: The Microbiological Assessment of Deep Carious Lesions After Step-wise Excavation and Diode Laser Cavity Disinfection .
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, shahenda gamal tawfik hamdy, internal resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: cebc-cu-2017-09-25
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Antibacterial Effect of Diode Laser
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: outcome assessor the assessor will not be blind about the type of intervention/control assessment methods. however it will not be allowed amongst the examiners to exchange any information throughout the entire study period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- disinfection the cavity with diode laser (Experimental): diode laser has antibacterial effect so can disinfect deep cavity and decrease the count of bacteria present after stepwise excavation
  Interventions: Device: diode laser
- no cavity disinfection (Placebo Comparator): placebo is used as no cavity disinfection will be done as after excavation the restoration will be placed .
  Interventions: Device: diode laser

INTERVENTIONS:
Device: diode laser — diode laser has antibacterial effect so can disinfect deep cavity and decrease the count of bacteria present after stepwise excavation

SUMMARY:
This study will be conducted to assess antibacterial effect of the diode laser in deep carious cavity after step wise excavation using the bacteriological assessment method.

DETAILED DESCRIPTION:
each patient should have at least two deep carious lesions The first clinical step in all teeth will be the opening of the cavity and the removal of undermined enamel . Caries at the lateral walls of the cavity and at the enamel-dentin junction was completely removed with excavators and/or round carbide burs at low speed. Subsequently, the central cariogenic biomasses and superficial part of the necrotic and demineralized dentin were removed. then excavation continued until the pulp exposure would occur with further excavation; thus, a layer of soft carious dentin was left on the cavity floor adjacent to the pulp wall.

A dentine samples will be then collected from the base of the cavity using sterile spoon excavator from the both groups for baseline bacteriological assessment and another sample will be taken after disinfection with diode laser in the intervention group .

In the two groups The remaining innermost layer of carious dentin are covered with calcium hydroxide The cavity was then sealed with restorative material (resin modified glass ionomer) after a 6 month period. This time was considered adequate for calcium hydroxide to exert its effect and for the pulp to respond with possible formation of tertiary dentin. The teeth were followed up every month and the integrity of the temporary restoration checked. After this interval of 6 months. After the rubber dam application, the temporary filling is removed samples are collected and the teeth are finally restored

ELIGIBILITY:
Inclusion Criteria:

1. Patients with at least two deep occlusal carious lesion .
2. 18 - 25years.
3. Males or Females.
4. Good oral hygiene.
5. Co-operative patients approving the trial and willing to sign a written consent.

Exclusion Criteria:

1. Pregnancy.
2. Systemic disease or severe medical complications.
3. Heavy smoking.
4. Xerostomia.
5. Lack of compliance.
6. Evidence of temporomandibular joint disorders.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2018-03-15 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
bacteriological count | 30 minute
  dentine samples will be taken before and after application of diode laser then bacteriological assessment will be done in the micro-lab